CLINICAL TRIAL: NCT02682355
Title: Optimizing Clinical Use of Polymyxin B: Teaching an Old Drug to Treat Superbugs
Brief Title: Optimizing Clinical Use of Polymyxin B
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Keith S. Kaye, MD, MPH, Project Director, Principal Investigator, Rutgers, The State University of New Jersey
Other Study IDs: R01AI119446-01 (NIH)
Record Dates: First submitted 2016-01-11; First posted 2016-02-15 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Pneumonia; Blood Stream Infection; Urinary Tract Infections; Respiratory Tract Infection (Including Tracheobronchitis); Sepsis
MeSH Terms: conditions — Pneumonia; Urinary Tract Infections; Respiratory Tract Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood and Respiratory cultures from infection site.
  * Urine Samples for Proteomic testing.
  * Blood Specimen for Pharmacokinetic/Pharmacodynamic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Patients receiving IV polymyxin B for treatment of bacteremia and/or urinary tract infection and/or respiratory tract infection (including tracheobronchitis) or sepsis

SUMMARY:
Polymyxin B is already being used extensively in the USA and other parts of the world; its use is likely to rapidly increase due to the greater burden of infections caused by MDR Gram-negative bacteria and the growing awareness of the limitations inherent in the clinical pharmacology of CMS/colistin. Cross resistance exists between the two polymyxins and thus both must be dosed optimally; but the recently generated scientifically-based dosage regimens for CMS/colistin cannot be extrapolated to polymyxin B. It is essential that an adequately powered study is conducted to define the clinical PK/PD/TD relationships of polymyxin B and identify, using next-generation proteomics, biomarkers for early detection of kidney injury. This will allow the development of scientifically-based dosage regimens for various categories of patients and an adaptive feedback control clinical tool for optimized dosing of polymyxin B in future individual patients.

DETAILED DESCRIPTION:
Multidrug-resistant (MDR) Gram-negative 'superbugs' are rapidly spreading around the world, and polymyxin B and colistin (polymyxin E) are often the only effective antibiotics. Since polymyxin B was released in the 1950s, its pharmacokinetics, pharmacodynamics, toxicodynamics (PK/PD/TD) have never been defined. Recent pharmacological research on polymyxins has predominantly focused on colistin methanesulfonate (CMS, an inactive prodrug of colistin) and demonstrates that CMS has significant limitations. Thus, polymyxin B is increasingly being viewed as the preferred polymyxin. Unfortunately, recently developed scientifically-based dosing recommendations for CMS cannot and should not be applied to polymyxin B, as the latter is administered as its active entity. Therefore, it is essential to determine the PK/PD/TD of polymyxin B in critically-ill patients, refine optimal dosage regimens, and develop the user-friendly adaptive feedback control (AFC) clinical tool.

The Specific Aims are:

1. To develop a population PK model for polymyxin B;
2. To investigate relationships between the PK of polymyxin B, duration of therapy and patient characteristics, with the development and timing of nephrotoxicity; and to use next-generation proteomics to identify the most predictive biomarker(s) of polymyxin B associated nephrotoxicity; and to develop the population PK/TD model;
3. To establish the relationships between polymyxin B PK, bacterial susceptibility and patient characteristics, with the probability of attaining and time to achieving clinical and bacteriological outcomes; and
4. To employ the models from Aims 1-3 and Monte Carlo simulation to develop scientifically-based dosage regimens of polymyxin B and to develop an AFC algorithm for future individual patients.

Research Design: Patients being treated with intravenous polymyxin B will be identified at three clinical sites in the USA and one in Singapore. Patients (n = 250) will have blood collected at various times surrounding a dose of polymyxin B between days 1 and 5 of therapy. Development of nephrotoxicity, clinical response, and bacteriological response will be examined. Total and free plasma concentrations of polymyxin B will be determined. Bacterial isolates will be examined for the emergence of polymyxin resistance. The relationships between polymyxin B PK, PD and TD end-points (e.g. clinical and bacteriological responses, development of toxicity and resistance) will be assessed using pharmacometric analyses. Finally, the obtained information will be used to apply Monte Carlo simulation to examine the impact of various patient characteristics and other factors on polymyxin B PK, PD and TD, in order to establish optimal dosage regimens and AFC algorithms for individual critically-ill patients.

Significance: No new antibiotics will be available for Gram-negative 'superbugs' for many years. This landmark multicenter study will provide essential information for optimizing polymyxin B use in critically-ill patients, while minimizing resistance and toxicity. This proposal aligns perfectly with the NIAID priority "To teach old drugs new tricks" and the recent Executive Order of the White House to combat antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of 18 years of age or older
2. Expectation of hospitalization and receipt of polymyxin B of ≥ 48 hours
3. Receipt of intravenous polymyxin B for treatment of bacteremia and/or urinary tract infection and/or respiratory tract infection (including tracheobronchitis) or sepsis
4. Provision of written informed consent by the patient or by the patient's health care proxy if the patient cannot give consent
5. Adequate venous access to enable collection of blood for determination of concentrations of polymyxin B and co-administered antibiotics

Exclusion Criteria:

1. Age <18 years
2. Currently incarcerated
3. Concomitant use of polymyxin B delivered directly into the respiratory tract
4. Cystic fibrosis
5. Known allergy to CMS/colistin or polymyxin B
6. Anticipated death within 48 h of commencing polymyxin B therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The human subjects involved in this study will be receiving intravenous polymyxin B as part of their routine clinical care because of infection due to bacteria resistant to all other first-line antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2016-02; Primary Completion 2022-05-31 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Polymyxin B plasma concentrations | 28 days after enrollment

SECONDARY OUTCOMES:
Changes in serum creatinine | 28 days after enrollment
Clinical response based on resolution of signs and symptoms of infection | 28 days after enrollment
Microbiologic response based on eradication of pathogens from blood and respiratory cultures | 28 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Keith S Kaye, MD, MPH, Principal Investigator — Rutgers University
Locations (6):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Columbia University Medical Center, New York, New York
  - New York Presbyterian-Weill Cornell Medical Center, New York, New York
- Brazil (2):
  - Hospital Sao Lucas da - PUC / RS, Porto Alegre
  - Hospital Moinhos de Vento, Porto Alegre
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT02682355/ICF_000.pdf